CLINICAL TRIAL: NCT06159426
Title: Electromyographic Response Control in the Application of Vojta Therapy in the Abdominal Muscles of Healthy Young Adults: Expert vs Non-expert Comparison
Brief Title: Expert vs. Non-expert Abdominal Electromyographic Control in Vojta Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Assistant professor doctor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NEUROUSAL04/2023
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Muscles
Keywords: Electromyography; Muscle Contraction; Expert Therapist; Outcome and Process Assessment; Health Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expert group (Experimental): The stimulation will be applied by an expert therapist.
  Interventions: Other: Vojta Therapy
- Non-expert group (Active Comparator): This group will receive the same stimulation as the expert group but in this case it will be applied by a therapist not specialized in therapy.
  Interventions: Other: Vojta Therapy

INTERVENTIONS:
Other: Vojta Therapy — The subject will be placed on a stretcher with the torso uncovered. Once the adhesive electrodes have been placed in the different recording areas on the anterior part of the trunk, a recording of the activity at rest will begin, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation in the contralateral side and, finally, one minute of rest.
  The therapy consists of the application of a stimulating pressure in the pectoral area in the pattern of the locomotion complex of reflex rolling in its first phase. For this, the subject will be placed in a supine position aligned with respect to the axial axis, with the arms along the body, the lower extremities in extension, and the head extended with a rotation of approximately 30º towards one side of the stimulation. The manual stimulation pressure will be exerted in the space between the 6th-7th or the 7th-8th rib under the mammillary line, with a force of about 2 kg.

SUMMARY:
Randomized clinical trial on a cohort of healthy subjects of legal age, of both sexes, recruited from the university community and who will be randomly distributed into two groups (expert therapist vs. non-expert therapist). The objective will be to determine if there are differences in the muscular activation produced on the stabilizing muscles of the trunk (external oblique and internal oblique) if it is applied by an expert therapist versus if it is applied by a therapist not specialized in therapy and to know the effects produced on the muscles studied after performing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Full cognitive capacity.

Exclusion Criteria:

* Subjects with neuro-muscular pathologies that affect the abdominal muscles, previous surgeries in the area or any chronic neurological or organic disorder that may alter the results.
* Vaccinated in the 10 days prior to the intervention
* Fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activity in abdominal muscles | Change from Baseline electromyographic activity at 7 minutes.
  The electromyographic activity of internal and external obliques in nanovolts will be collected before, during and after the intervention.

SECONDARY OUTCOMES:
Date of birth | Baseline
  It will be registered at the beginning of the study in order to calculate the age of the participant.
Sex | Baseline
  It will be registered at the beginning of the study.
Height | Baseline
  It will be registered at the beginning of the study in centimeters.
Weight | Baseline
  It will be registered at the beginning of the study in kilograms.

IPD SHARING:
Plan to Share IPD: Undecided